CLINICAL TRIAL: NCT04339738
Title: A Multicenter Phase II Trial of Paclitaxel With and Without Nivolumab in Taxane Naive, and Nivolumab and Cabozantinib in Taxane Pretreated Subjects With Angiosarcoma
Brief Title: Testing the Addition of Nivolumab to Chemotherapy in Treatment of Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-02153; NCI-2020-02153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A091902 (Other: Alliance for Clinical Trials in Oncology); A091902 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Skin Angiosarcoma; Skin Radiation-Related Angiosarcoma; Visceral Angiosarcoma
MeSH Terms: interventions — Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy; Nivolumab; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (nivolumab, paclitaxel) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and paclitaxel IV over 1 hour on days 1, 8, and 15. Cycles repeat every 4 weeks for up to 2 years (24 months) for patients who achieve CR, PR or SD on immunotherapy/nivolumab, or in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood at baseline and on study, CT scan, spiral CT, or MRI, or FDG-PET scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Cycles repeat every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood at baseline and on study, CT scan, spiral CT, or MRI, or FDG-PET scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (nivolumab, cabozantinib S-malate) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and cabozantinib S-malate PO daily. Cycles repeat every 4 weeks for up to 2 years (24 months) for patients who achieve CR, PR or SD on immunotherapy/nivolumab, or in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood at baseline and on study, CT scan, spiral CT, or MRI, or FDG-PET scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm III (nivolumab, cabozantinib S-malate)
Procedure: Computed Tomography — Undergo CT, spiral CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm I (nivolumab, paclitaxel); Arm III (nivolumab, cabozantinib S-malate)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (nivolumab, paclitaxel); Arm II (paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well paclitaxel with and without nivolumab works in treating patients with soft tissue sarcoma that have not received taxane drugs, and how well nivolumab and cabozantinib work in treating taxane pretreated patients with soft tissue sarcoma. Nivolumab works through the body's immune system to help the immune system act against tumor cells. Chemotherapy drugs, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This trial is being done to see if the combination of nivolumab and paclitaxel or cabozantinib can shrink soft tissue sarcoma and possibly prevent it from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression free survival (PFS) for paclitaxel with and without nivolumab in subjects with taxane naive angiosarcoma.

II. To determine the overall response rate (ORR) of nivolumab in combination with cabozantinib S-malate (cabozantinib) in patients with taxane pre-treated angiosarcoma.

SECONDARY OBJECTIVES:

I. To determine the ORR of paclitaxel in combination with nivolumab. II. To determine clinical activity of the addition of nivolumab to paclitaxel or cabozantinib in subjects with angiosarcoma by determination of overall survival (OS) for each combination.

III. To determine clinical activity of the addition of nivolumab to cabozantinib in subjects with taxane pre-treated angiosarcoma by determination of progression free survival (PFS) at 6 months by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria.

IV. To assess toxicity of the concurrent nivolumab-paclitaxel and nivolumab-cabozantinib combinations in subjects with angiosarcoma based on National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.

V. To measure symptomatic adverse events (AE) for patients via Patient Reported Outcome (PRO)-CTCAE, Functional Assessment of Cancer Therapy General (FACT-G) questionnaire, and Linear Analogue Self-Assessment (LASA).

OUTLINE: Patients who have not previously received a taxane are randomized to Arm I or Arm II. Patients who have previously received a taxane are assigned to Arm III.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and paclitaxel IV over 1 hour on days 1, 8, and 15. Cycles repeat every 4 weeks for up to 2 years (24 months) for patients who achieve complete response (CR), partial response (PR) or stable disease (SD) on immunotherapy/nivolumab, or in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Cycles repeat every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm III.

ARM III (EFFECTIVE OF 10/28/2021, NEW PATIENT ACCRUAL PERMANENTLY CLOSED): Patients receive nivolumab IV over 30 minutes on day 1 and cabozantinib orally (PO) daily. Cycles repeat every 4 weeks for up to 2 years (24 months) for patients who achieve CR, PR or SD on immunotherapy/nivolumab, or in the absence of disease progression or unacceptable toxicity.

Patients also undergo collection of blood at baseline and on study, computed tomography (CT) scan, spiral CT, or magnetic resonance imaging (MRI), or FDG-positron emission tomography (FDG-PET) scan throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cutaneous or visceral angiosarcoma, where curative treatment is either not possible or curative modality therapy is declined by the subject. Note: If a subject declines curative modality therapy, the reason must be documented (e.g. excessive morbidity to necessary surgery)

  * Note: Radiation induced angiosarcomas are permitted

    * All local diagnostic slides AND 5 x 4-6 micron unstained slides from diagnostic tumor tissue should be available for retrospective central pathology review
* Must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Per RECIST v1.1, clinical lesions will only be considered measurable when they are superficial and >= 10 mm diameter as assessed using calipers or ruler (e.g. skin nodules). For the case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is required. When lesions can be evaluated by both clinical exam and imagining, imaging evaluation should be undertaken since it is more objective and may also be reviewed at the end of the study. The same method of measurement should be used throughout the study, preferably performed by the same investigator. Areas previously radiated must have demonstrated disease progression at some point over the past 6 months and growth must be subsequent to the last line of anti-cancer directed therapy (e.g. chemotherapy, radiation therapy, surgery)
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 3 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Prior Treatment

  * Patient must have completed all prior cancer directed therapies (including investigational) >= 7 days prior to cycle 1 day 1

    * Exception: prostate patients who are allowed to concurrently receive androgen suppression therapy
    * Note: Radiation therapy must be completed >= 7 days of day 1 of study treatment, and must not be expected to significantly impact blood count recovery
  * There is no limit to overall number of prior lines of therapy
  * No prior PD-1 inhibitor or PD-L1 inhibitor therapy is permitted
  * No prior administration of VEGF TKI therapy is permitted
  * Recovery to baseline or' =< grade 1 CTCAE version 5.0 from toxicity related to any prior treatment, unless adverse events are clinically non-significant and/or stable on supportive therapy, with the exception of fatigue (which should be =< grade 2) or alopecia. Note: Patients should be expected to have experienced any nadir and have adequate blood count recovery prior to cycle 1 day 1
* Taxane Naive Patients Only: No prior exposure to taxane therapy of any duration for angiosarcoma
* Taxane Pre-treated Patients Only (Effective 10/28/2021, new patient accrual to Arm 3 was permanently closed): Prior taxane therapy is allowed at any point prior to registration as long as prior treatment eligibility criteria are met prior to cycle 1 day 1
* No major surgery (except the diagnostic biopsy) =< 28 days of study registration. Procedures such as thoracentesis, paracentesis, percutaneous biopsy, Lasik eye surgery are not considered major surgery. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Calculated (Calc.) creatinine clearance >= 30 mL/min (per Cockcroft-Gault)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * For patients with documented/suspected Gilbert's disease, bilirubin =< 3 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)

  * For patients with significant hepatic metastases, ALT and AST =< 5 x ULN. No clinically active or chronic liver disease resulting in moderate/severe hepatic impairment (Child-Pugh class B or C), ascites, coagulopathy or bleeding due to liver dysfunction
* Urine protein:creatinine (UPC) ratio < 1 or urine protein =< 1+ (Only for Arm 3 Taxane pre-treated and crossover patients)
* No uncontrolled central nervous system (CNS) metastases. Patients with history of CNS metastasis will be allowed as long as the metastatic sites were adequately treated as demonstrated by clinical and radiographic improvement, and the patient has recovered from the intervention (no residual adverse events > CTCAE grade 1), and the patient has remained without recurrence of new or worsening CNS symptoms for a period of 28 days prior to registration. Treated CNS metastasis (mets) should have no ongoing requirement for steroids, and no evidence of hemorrhage after treatment for at least 28 days prior to registration
* No uncontrolled intercurrent illness that would put the patient at undue risk by participation in the study, in the opinion of the investigator
* No history of syncope of cardiovascular etiology, uncontrolled cardiac arrhythmia, history of Mobitz II second degree or third degree heart block without a permanent pacemaker in place, myocardial ischemia or infarction, severe or unstable angina, New York Heart Association (NYHA) class II to IV heart failure, or stroke/transient ischemic attack (TIA) within the past 3 months
* No thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 1 month before randomization. Subjects with a diagnosis of incidental, subsegmental pulmonary embolism (PE) or deep vein thrombosis (DVT) within 6 months are allowed if stable, asymptomatic, and treated with low molecular weight heparin (LMWH) for at least 2 weeks before first dose. Iatrogenic arterial embolization procedures such as tumor arterial embolization or splenic artery embolization are allowed
* Patients with a requirement for steroid treatment or other immunosuppressive treatment: Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Active autoimmune disease requiring systemic treatment (i.e. disease modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. These include but are not limited to patients with a history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease

  * Note: Patients are permitted to enroll if they have vitiligo; type I diabetes mellitus; hypothyroidism, pituitary or adrenal insufficiency requiring only hormone replacement; psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* No planned palliative procedures for alleviation of pain such as radiation therapy or surgery
* No untreated or impending spinal cord compression or evidence of spinal metastases with a risk of impending fracture or spinal cord compression
* No known or suspected contraindications or hypersensitivity to paclitaxel, cabozantinib or nivolumab or to any of the excipients
* Disorders associated with a high risk of perforation or fistula formation: active inflammatory bowel disease, active diverticulitis, active cholecystitis, active symptomatic cholangitis or active appendicitis, active acute pancreatitis or active acute obstruction of the pancreatic or biliary duct, or active gastric outlet obstruction; abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before randomization. Note: Complete healing of an intra-abdominal abscess must be confirmed before randomization
* No clinically significant hematuria, hematemesis, or hemoptysis, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 3 months before randomization
* No lesions invading major pulmonary blood vessels
* No other clinically significant disorders: uncompensated/symptomatic hypothyroidism; requirements for hemodialysis or peritoneal dialysis; history of solid organ transplantation
* Serious non-healing wounds unrelated to cancer are excluded

  * Note: Wounds that are cutaneous angiosarcoma are allowed
* Chronic concomitant treatment with strong inhibitors and inducers of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors and inducers must discontinue the drug 7 days and 14 days, respectively prior to registration on the study
* Taxane Naive Patients Only: No clinically significant neuropathy (grade >= 2 per NCI CTCAE v5.0)
* Taxane Pre-treated only (Effective 10/28/2021, new patient accrual to Arm 3 was permanently closed):

  * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose. Subjects with a diagnosis of DVT within 6 months are allowed if stable and treated with LMWH for at least 2 weeks before first dose
  * No history of clinically significant coagulopathy
  * No uncontrolled hypertension, defined as systolic blood pressure of > 140 mmHg or diastolic pressure > 90 mmHg on anti-hypertensive medications
  * No known or suspected gastrointestinal disorder affecting absorption of oral medications (for patients getting cabozantinib)
* No clinical, laboratory or radiographic evidence of an active bacterial, fungal, or viral infection requiring treatment at the time of registration. No concurrent use of parenteral (IV) antibiotics is permitted. Oral antibiotics administered for a defined course with expectation of resolution of infection are permitted at the discretion of the investigator
* No use of ongoing systemic steroid therapy within 7 days prior to study registration. Dose equivalence of prednisone 10mg daily or less is permitted
* Taxane Pre-treated only:

  * No current use of aspirin (> 81 mg/day), or any other antiplatelet agents
  * Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin inhibitors, and factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel) is not permitted. Low-dose (prophylactic) low molecular weight heparins (LMWH) are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects with no known brain metastases, no clinically significant hemorrhage, or no complications from a thromboembolic event on the anticoagulation regimen, and who have been on a stable dose of LMWH for at least 2 weeks before first dose
* Patients must be able to speak and comprehend English or Spanish in order to complete the mandatory patient-completed measures
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 3 days prior to re-registration is required
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Age >= 18 years
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): ECOG performance status 0-1
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Prior Treatment

  * Patient must have completed all prior treatments (including investigational Arm 2 paclitaxel) >= 28 days prior to cycle 1 day 1

    * Exception: prostate patients who are allowed to concurrently receive androgen suppression therapy
    * Note: Re-registration is only permitted after progression on Arm 2
  * No prior PD-1 inhibitor or PD-L1 inhibitor therapy is permitted
  * Recovery to baseline, or =< grade 1 CTCAE version 5.0 from toxicity related to any prior treatment, unless adverse events are clinically non-significant and/or stable on supportive therapy, with the exception of fatigue (which should be =< grade 2) or alopecia. Note: Patients should be expected to have experienced any nadir and have adequate blood count recovery prior to cycle 1 day 1
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No major surgery (except the diagnostic biopsy) =< 28 days of study re-registration. Procedures such as thoracentesis, paracentesis, percutaneous biopsy, Lasik eye surgery are not considered major surgery. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Absolute neutrophil count (ANC) >= 1,500/mm^3
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Platelet count >= 100,000/mm^3
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Hemoglobin >= 9.0 g/dL
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Calc. creatinine clearance >= 30 mL/min (per Cockcroft-Gault)
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * For patients with documented/suspected Gilbert's disease, bilirubin =< 3 x ULN
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): AST/ALT =< 2.5 x upper limit of normal (ULN)

  * For patients with significant hepatic metastases, ALT and AST =< 5 x ULN. No clinically active or chronic liver disease resulting in moderate/severe hepatic impairment (Child-Pugh class B or C), ascites, coagulopathy or bleeding due to liver dysfunction
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): UPC ratio < 1 or urine protein =< 1+
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No uncontrolled CNS metastases. Patients with history of CNS metastasis will be allowed as long as the metastatic sites were adequately treated as demonstrated by clinical and radiographic improvement, and the patient has recovered from the intervention (no residual adverse events > CTCAE grade 1), and the patient has remained without recurrence of new or worsening CNS symptoms for a period of 28 days prior to registration. Treated CNS mets should have no ongoing requirement for steroids, and no evidence of hemorrhage after treatment for at least 28 days prior to registration
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No uncontrolled intercurrent illness that would put the patient at undue risk by participation in the study, in the opinion of the investigator
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No history of syncope of cardiovascular etiology, uncontrolled cardiac arrhythmia, History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place, myocardial ischemia or infarction, severe or unstable angina, New York Heart Association (NYHA) class II to IV heart failure, or stroke/transient ischemic attack (TIA) within the past 3 months
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 1 month before randomization. Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with LMWH for at least 2 weeks before first dose. Iatrogenic arterial embolization procedures such as tumor arterial embolization or splenic artery embolization are allowed
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Patients with a requirement for steroid treatment or other immunosuppressive treatment: Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): Active autoimmune disease requiring systemic treatment (i.e. disease modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. These include but are not limited to patients with a history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease

  * Note: Patients are permitted to enroll if they have vitiligo; type I diabetes mellitus; hypothyroidism, pituitary or adrenal insufficiency requiring only hormone replacement; psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No planned palliative procedures for alleviation of pain such as radiation therapy or surgery
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No untreated or impending spinal cord compression or evidence of spinal metastases with a risk of impending fracture or spinal cord compression
* Re-Registration Eligibility Criteria (upon progression on Arm 2 only): No known or suspected contraindications or hypersensitivity to cabozantinib or nivolumab or to any of the exc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in taxane naive patients with angiosarcoma | From registration (randomization) to either progression or death (without progression), assessed up to 3 years
  Will compare the PFS in taxane naive angiosarcoma patients receiving either (1) paclitaxel + nivolumab compared to (2) paclitaxel alone.
Overall response rate (ORR) in angiosarcoma patients who have had prior taxane | Up to 3 years
  Will compare the overall response rate (ORR) of nivolumab + cabozantinib in patients with angiosarcoma who have had prior taxanes to historical control of VEGF inhibitors alone.

SECONDARY OUTCOMES:
ORR in the nivolumab + paclitaxel | Up to 3 years
  Will be estimated by dividing the number of evaluable patients that achieve a confirmed response by the total number of evaluable patients in the nivolumab + paclitaxel combination arm. Additionally a 95% confidence interval will be constructed utilizing properties of the binomial distribution.
Overall survival in each of the 2 combination arms | From study enrollment until death due to any cause, assessed up to 3 years
  Will be evaluated using the Kaplan-Meier method in order to determine the median survival rate. This median survival rate will be calculated for each of the 2 combination arms (i.e. nivolumab + paclitaxel and nivolumab + cabozantinib).
PFS rate | At 6 months
Incidence of adverse events | Up to 3 years
  Maximum grade adverse events will be summarized by treatment arm in a tabular setting. This will be done both with and without regard to the assigned attribution of each adverse event.
Patient-reported outcomes (PRO) | Up to 3 years
  Will be assessed via PRO-Common Terminology Criteria for Adverse Events (CTCAE). In order to evaluate this endpoint we will calculate the proportion of patients that report a grade 3+ event along with a 95% confidence interval based on the properties of the binomial distribution. Any other analyses with these data will be done in an exploratory and hypothesis generating manner.

CONTACTS AND LOCATIONS:
Overall Officials: Juneko E Grilley-Olson, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (171):
- United States (170):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- FHP Health Center-Guam, Tamuning, Guam

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT04339738/ICF_000.pdf